CLINICAL TRIAL: NCT02040753
Title: The Effect of Repeated Lifestyle Intervention on Weight Loss Maintenance
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Ubberup Folk High School (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Associate Professor, University of Copenhagen
Other Study IDs: UBBERUP1
Record Dates: First submitted 2013-11-21; First posted 2014-01-20 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Overweight
Keywords: Lifestyle intervention; Change of body composition; Physical activity; Weight loss maintenance
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intensive Lifestyle Intervention: Former participants of intensive lifestyle intervention at Ubberup Folk High School.
  Interventions: Behavioral: Intensive Lifestyle Intervention

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — Intensive Lifestyle intervention at Ubberup Folk High School for 10-14 weeks. Daily exercise for 1-3hrs. Calorie restriction. Education within Nutrition, exercise and healthy living in general.

SUMMARY:
In Denmark and the western world, there is an increasing prevalence of obesity probably due to a combination of inadequate daily physical activity and a high energy intake. One approach to achieve weight loss and change life style is to participate in an intensive supervised prolonged life style modification course. The immediate effect is often positive, but over time the overall effect is limited as the majority will not maintain weight loss and a changed life style.

In this study we will analyse the results of the intensive lifestyle intervention as it has been practised at Ubberup Folk High School over the last 13 years. As some people have several stays at Ubberup Folk High School we want to we have a special interest in the effect of repeated lifestyle intervention.

Research question:

What is the effect of several lifestyle interventions on weight loss maintenance?

The study design is retrospective and descriptive and will be based on a lifestyle intervention, as it has practiced in a real life setting at Ubberup folk high school.

ELIGIBILITY:
Inclusion Criteria:

* Former participants of the intensive lifestyle intervention at Ubberup Folk High School.

Exclusion Criteria:

* Gastric bypass surgery or banding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Former participants of Ubberup Folk High School.
Sampling Method: Non-Probability Sample
Enrollment: 2120 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in total body weight | Before intervention, after intervention (after 10-14 weeks) and follow up measurements after 1-13 years depending on when the lifestyle intervention took place

SECONDARY OUTCOMES:
Change in body composition | Before intervention, after intervention (after 10-14 weeks) and follow up measurements after 1-13 years depending on when the lifestyle intervention took place
  Measured by bio-impedance.

CONTACTS AND LOCATIONS:
Overall Officials: Jørn W Helge, PhD, Principal Investigator — University of Copenhagen, Department of Biomedical Sciences
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen, Denmark

REFERENCES:
- [Background] Karlsen TI, Sohagen M, Hjelmesaeth J. Predictors of weight loss after an intensive lifestyle intervention program in obese patients: a 1-year prospective cohort study. Health Qual Life Outcomes. 2013 Oct 3;11:165. doi: 10.1186/1477-7525-11-165. PMID 24090083
- [Background] McCormack SE, McCarthy MA, Harrington SG, Farilla L, Hrovat MI, Systrom DM, Thomas BJ, Torriani M, McInnis K, Grinspoon SK, Fleischman A. Effects of exercise and lifestyle modification on fitness, insulin resistance, skeletal muscle oxidative phosphorylation and intramyocellular lipid content in obese children and adolescents. Pediatr Obes. 2014 Aug;9(4):281-91. doi: 10.1111/j.2047-6310.2013.00180.x. Epub 2013 Jun 25. PMID 23801526
- [Background] Danielsen KK, Svendsen M, Maehlum S, Sundgot-Borgen J. Changes in body composition, cardiovascular disease risk factors, and eating behavior after an intensive lifestyle intervention with high volume of physical activity in severely obese subjects: a prospective clinical controlled trial. J Obes. 2013;2013:325464. doi: 10.1155/2013/325464. Epub 2013 Apr 22. PMID 23710347
- [Background] Bruun JM, Helge JW, Richelsen B, Stallknecht B. Diet and exercise reduce low-grade inflammation and macrophage infiltration in adipose tissue but not in skeletal muscle in severely obese subjects. Am J Physiol Endocrinol Metab. 2006 May;290(5):E961-7. doi: 10.1152/ajpendo.00506.2005. Epub 2005 Dec 13. PMID 16352667
- [Background] Pedersen JO, Zimmermann E, Stallknecht BM, Bruun JM, Kroustrup JP, Larsen JF, Helge JW. [Lifestyle intervention in the treatment of severe obesity]. Ugeskr Laeger. 2006 Jan 9;168(2):167-72. Danish. PMID 16403343
- [Background] Bruun JM, Stallknecht B, Helge JW, Richelsen B. Interleukin-18 in plasma and adipose tissue: effects of obesity, insulin resistance, and weight loss. Eur J Endocrinol. 2007 Oct;157(4):465-71. doi: 10.1530/EJE-07-0206. PMID 17893261
- [Background] Christiansen T, Bruun JM, Madsen EL, Richelsen B. Weight loss maintenance in severely obese adults after an intensive lifestyle intervention: 2- to 4-year follow-up. Obesity (Silver Spring). 2007 Feb;15(2):413-20. doi: 10.1038/oby.2007.530. PMID 17299115
- [Derived] Dandanell S, Skovborg C, Praest CB, Kristensen KB, Nielsen MG, Lionett S, Jorgensen SD, Vigelso A, Dela F, Helge JW. Maintaining a clinical weight loss after intensive lifestyle intervention is the key to cardiometabolic health. Obes Res Clin Pract. 2017 Jul-Aug;11(4):489-498. doi: 10.1016/j.orcp.2016.09.009. Epub 2016 Oct 5. PMID 27720417